CLINICAL TRIAL: NCT02171390
Title: Phase 4 Study That Evaluates the Presence of Endothelial Dysfunction, Inflammation and Insulin Resistance in Male Subjects With Hypogonadotrophic Hypogonadism and Effects of Two Different Testosterone Replacement Regiments on These Parameters.
Brief Title: Endothelial Dysfunction, Inflammation and Insulin Resistance in Congenital Hypogonadism and Effect of Testosteron Replacement Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Alper Sonmez, Associate Professor in Medicine, Gulhane School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GSM-042014
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-03

CONDITIONS: Hypogonadotrophic Hypogonadism
Keywords: Hypogonadism; Endothelial dysfunction; Insulin resistance; Inflammation; Testosterone replacement therapy
MeSH Terms: conditions — Hypogonadism; Insulin Resistance; Inflammation | interventions — Testosterone; Injections; Adenosine Monophosphate; Testosterone Propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily testosterone transdermal gel (Active Comparator)
  Interventions: Drug: Testosteron 50 mg transdermal gel
- Injectable Testosterone esters (Active Comparator): Testosteron 250mg injection per 3-4 weeks for 6 months
  Interventions: Drug: Testosterone 250mg injection

INTERVENTIONS:
Drug: Testosterone 250mg injection — The testosterone 250mg ester intramuscular injections performed in three weeks
  Other Names: Sustanon 250 mg amp.
  Arms: Injectable Testosterone esters
Drug: Testosteron 50 mg transdermal gel — 50mg testosterone gel implemented on every night
  Other Names: Testogel 50mg transdermal gel
  Arms: Daily testosterone transdermal gel

SUMMARY:
The study searched for answers to two questions

1. Is there endothelial dysfunction, inflammation and insulin resistance in patients with congenital hypogonadotropic hypogonadism?
2. What is the effect of testosterone replacement therapy on endothelial dysfunction, inflammation and insulin resistance?

ELIGIBILITY:
Inclusion Criteria:

* Men
* Treatment naive
* Hypogonadotrophic hypogonadism

Exclusion Criteria:

* Previous history of androgen replacement
* Chronic metabolic disorders

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2008-08; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The alterations in the measures for endothelial functions | 6 months
  The alterations in Endothelial functions are determined by measuring plasma asymmetric dimethylarginine (ADMA) levels, as a surrogate. ADMA measurement is performed by ELISA kit (Immunodiagnostic, Bernheim, Germany)(Catalog Number 7828) with a minimal detection limit of 0.05µmol/L.
The alterations in the measures of inflammation | 6 months
  The alterations in the measures of inflammation are determined by measuring plasma TWEAK levels. ELISA kit (Bender MedSystems, Lot Nr.BMS2006INST, Vienna, Austria) was used.
The alterations in the measures of insulin resistance | 6 months.
  The alterations in insulin sensitivity are estimated by using the homeostasis model assessment (HOMA) index by the formula, HOMA = (insulin x glucose)/405.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine Department of Endocrinology and Metabolism, Ankara, NonUS, Turkey (Türkiye)